CLINICAL TRIAL: NCT00694603
Title: A Phase II Trial of Cetuximab (c225) as Therapy for Recurrent Non-Small Cell Lung Cancer in Patients Who Have Received Prior Therapy With Tyrosine Kinase Inhibitor Directed Against the EGFR Pathway
Brief Title: Cetuximab as Therapy for Recurrent Non-Small Cell Lung Cancer Patients Who Have Received Prior Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Lecia V. Sequist (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Unity Health Toronto (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Lecia V. Sequist, Overall PI, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-026
Record Dates: First submitted 2007-12-28; First posted 2008-06-10 (Estimated); Results first posted 2012-09-06 (Estimated); Last update posted 2012-09-06 (Estimated); Status verified 2012-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: cetuximab; tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab (Experimental): 400mg/m2 IV x 1 and then 250mg/m2 IV weekly
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Given intravenously once per week.
  Other Names: Erbitux

SUMMARY:
The purpose of this research study is to find out how well cetuximab works in treating NSCLC in patients who have been previously treated with a class of drug called tyrosine kinase inhibitor (TKI). Cetuximab is a protein that is designed to block a substance in cancer cells called "epidermal growth factor receptor" or EGFR. EGFR helps cancer cells grow.

DETAILED DESCRIPTION:
* Participants on this study will receive cetuximab by infusion intravenously once per week and may continue to receive weekly cetuximab infusions until their disease progresses or they experience unacceptable side effects.
* The following will be performed every 4 weeks while they are receiving study treatments: Physical examination; performance status; and blood work. A CT scan of the chest and upper abdomen will be performed every 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage IIIB or IV recurrent or progressive NSCLC
* Patients must have progressed while receiving treatment with a tyrosine kinase inhibitor targeting the EGFR pathway
* Measurable disease, as defined by RECIST criteria
* Patients must have a suitable frozen or paraffin-embedded tissue sample available for EGFR mutational analysis. Prior EGFR mutational analyses are allowable
* Patients with asymptomatic brain metastasis are eligible; however, they must have completed radiotherapy/radiosurgery at least 3 weeks prior to enrollment and be clinically stable
* ECOG Performance Status 0-2
* 18 years of age or older
* Negative pregnancy test within 7 days of treatment or be categorized as not of child-bearing potential
* Bone marrow function, renal function, hepatic function as outlined in protocol

Exclusion Criteria:

* Women who are pregnant of breastfeeding
* Active concurrent malignancy
* Major thoracic or abdominal surgery within 30 days prior to the first infusion of cetuximab
* Significant history of uncontrolled cardiac disease
* Uncontrolled seizure disorder, or active neurological disease
* Prior severe infusion reactions to a monoclonal antibody
* Prior chemotherapy regimen within 21 days prior to study entry
* Any EGFR tyrosine kinase inhibitor within 14 days of study entry
* Radiation therapy within 14 days prior to the first infusion of cetuximab
* Acute hepatitis or known HIV
* Active or uncontrolled infection
* Any concurrent chemotherapy or any other investigational agent(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lecia Sequist, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Neal JW, Heist RS, Fidias P, Temel JS, Huberman M, Marcoux JP, Muzikansky A, Lynch TJ, Sequist LV. Cetuximab monotherapy in patients with advanced non-small cell lung cancer after prior epidermal growth factor receptor tyrosine kinase inhibitor therapy. J Thorac Oncol. 2010 Nov;5(11):1855-8. doi: 10.1097/JTO.0b013e3181f0bee0. PMID 20975380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patients to this multicenter, single-arm, phase II clinical trial with ECOG PS 0 to 2 and advanced NSCLC who were previously treated with erlotinib or gefitinib. Patients with asymptomatic, stable CNS metastases were eligible. 18 eligible patients were enrolled in the first stage of the trial between October 2006 and March 2009.
Pre-assignment Details: All patients were required to have an available tissue sample for EGFR mutation testing, which was performed centrally at a CLIA-certified laboratory.
Groups:
- Cetuximab: Patients received intravenous cetuximab, 400 mg/m2, followed by weekly infusions of 250 mg/m2. Four weekly treatments constituted one cycle.
Period: Overall Study
Arm/Group | Cetuximab
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Response Rate by CT Scan Using RECIST Criteria
Time Frame: 8 weeks
Population: The trial used a Simon two-stage design, which enrolled 18 pts in the first stage and was to proceed to enroll an additional 28 evaluable patients if 1 or more response was observed in the first group. This design provided a 57% chance of early termination if the true response rate was <3%. PFSand OS were calculated using the Kaplan-Meier method.
Measure: Number; unit: participants
Arm/Group | Cetuximab
Number analyzed (Participants) | 18
participants | 0

2. Secondary Outcome: Progression-free Survival
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab
Number analyzed (Participants) | 18
months | 1.8 [1.6 to 5.4]

ADVERSE EVENTS:
Arm/Group | Cetuximab
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 15/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=18)
interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
headache (Nervous system disorders) | 1
chest pain (Cardiac disorders) | 1
wheezing (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=18)
rash (Skin and subcutaneous tissue disorders) | 8
nausea (Gastrointestinal disorders) | 3
fatigue (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No